CLINICAL TRIAL: NCT01464892
Title: Rescripting With vs. Without Prior Stabilization in PTSD Following Early Chronic Interpersonal Trauma
Brief Title: Imagery Rescripting in the Treatment of Post Traumatic Stress Disorder (PTSD) Following Early Chronic Interpersonal Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Responsible Party: Principal Investigator, Mrs. M. Kindt, Professor of Experimental and Clinical Psychology, University of Amsterdam
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-KP-877
Record Dates: First submitted 2011-10-25; First posted 2011-11-04 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Imagery rescripting; Imagery rescripting and reprocessing therapy; Skills Training in affective and interpersonal regulation; Post-traumatic Stress Disorder; Childhood abuse; Childhood sexual abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Imagery Rescripting (Experimental)
  Interventions: Behavioral: Imagery Rescripting and Reprocessing Therapy
- STAIR plus Imagery Rescripting (Active Comparator)
  Interventions: Behavioral: STAIR + Imagery Rescripting
- Wait-list control (No Intervention): Participants from this arm are randomized to the two active conditions after 8 weeks of waiting.

INTERVENTIONS:
Behavioral: Imagery Rescripting and Reprocessing Therapy — This intervention is comprised of 16 sessions (twice a week) of trauma-focused imagery rescripting
  Other Names: IRRT
  Arms: Imagery Rescripting
Behavioral: STAIR + Imagery Rescripting — A two-phased treatment. Phase 1 is comprised of 8 (weekly) sessions of Skills Training in Affective and Interpersonal Skills (STAIR). Phase 2 consists of 16 sessions (twice weekly) of trauma-focused imagery rescripting.
  Arms: STAIR plus Imagery Rescripting

SUMMARY:
Imagery Rescripting (IR)is a promising treatment for PTSD in adult survivors of early, chronic, interpersonal trauma (e.g. Smucker & Dancu, 1999). So far, this protocol has not been investigated within a controlled setting with patients with PTSD following early, chronic, interpersonal trauma. The aim of the proposed study is to 1. investigate the efficacy of Imagery Rescripting and 2. check whether the efficacy of Imagery Rescripting can be improved by adding a stabilization phase (Skills training in affective and interpersonal regulation, STAIR) prior to this treatment. In a randomized controlled trial three conditions will be compared:

1. Imagery Rescripting
2. STAIR + Imagery Rescripting
3. Wait-list control

ELIGIBILITY:
Inclusion Criteria:

* a full diagnosis of post-traumatic stress disorder (PTSD) according to DSM-IV
* having experienced repeated or chronic interpersonal trauma by care-takers or authority figures before the age of 15
* between the age of 18 and 65 years
* sufficient fluency of Dutch to complete treatment and research-protocol
* participants using prescribed anti-depressant medication are required to be on a stable dose for at least 6 weeks before the beginning of treatment and remain on this dose throughout the treatment

Exclusion Criteria:

* psychosis
* bipolar disorder
* significant cognitive impairment
* substance dependence
* current use of benzodiazepines
* severe suicidal ideation or life-threatening automutilation
* current trauma or threat
* unstable living circumstances
* antisocial personality disorder
* primary diagnosis of borderline personality disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinician-Administered PTSD Scale (CAPS) at 8 weeks | baseline and 8 weeks
  comparison STAIR vs ImRs vs WL
Change from Baseline in Posttraumatic Diagnostic Scale (PDS) at 8 weeks | baseline and 8 weeks
  comparison STAIR vs ImRs vs WL

SECONDARY OUTCOMES:
Change from Baseline in Beck Depression Inventory (BDI)at 8 weeks | baseline and 8 weeks
Change from Baseline in Buss-Durkee Hostility Inventory (BDHI)at 8 weeks | baseline and 8 weeks
Change from Baseline in Inventory of Interpersonal Problems (IIP)at 8 weeks | baseline and 8 weeks
Change from Baseline in Dissociation Questionnaire (DIS-Q)at 8 weeks | baseline and 8 weeks
Change from Baseline in WHO-Quality of Life(WHO-QL)at 8 weeks | baseline and 8 weeks
Change from Baseline in Difficulties in Emotion Regulation Scale (DERS)at 8 weeks | baseline and 8 weeks
Change from Baseline in Structured Clinical Interview - Axis I (SCID-1)at 8 weeks | baseline and 8 weeks
Posttreatment: Change from Baseline in Clinician-Administered PTSD Scale (CAPS)at 8 weeks (ImRs) vs 16 weeks (STAIR/ImRs; WL/ImRs) vs 24 weeks (WL/STAIR/ImRs) | baseline and max.24 weeks (depending on condition)
12-week follow-up: Change from Baseline in Clinician-Administered PTSD Scale (CAPS) at 20 weeks (ImRs) vs 28 weeks (STAIR/ImRs; WL/ImRs) vs. 36 weeks (WL/STAIR/ImRs). | baseline and max. 36 weeks (depending on condition)
Post-treatment: Change from Baseline in Posttraumatic Diagnostic Scale (PDS) at 8 weeks (ImRs) vs 16 weeks (STAIR/ImRs; WL/ImRs) vs. 24 weeks (WL/STAIR/ImRs) | baseline and max.24 weeks (depending on condition)
12-week fu: Change from Baseline in Posttraumatic Diagnostic Scale (PDS) at 20 weeks (ImRs) vs 28 weeks (STAIR/ImRs; WL/ImRs) vs. 36 weeks (WL/STAIR)./ImRs). | baseline and max. 36 weeks (depending on condition)
Post-treatment: Change from Baseline in Beck Depression Inventory (BDI) at 8 weeks (ImRs) vs 16 weeks (STAIR/ImRs; WL/ImRs) vs. 24 weeks (WL/STAIR). | baseline and max 24 weeks (depending on condition)
Change from Baseline in Beck Depression Inventory (BDI) at 20 weeks (ImRs) vs 12-week-fu: 8 weeks (STAIR/ImRs; WL/ImRs) vs. 36 weeks (WL/STAIR). | baseline and max 36 weeks (depending on condition)
Post-treatment: Change from Baseline in Buss-Durkee Hostility Inventory (BDHI) at 8 weeks (ImRs) vs 16 weeks (STAIR/ImRs; WL/ImRs) vs. 24 weeks (WL/STAIR | baseline and max 24 weeks (depending on condition)
12-week FU: Change from Baseline in Buss-Durkee Hostility Inventory (BDHI) at 20 weeks (ImRs) vs 28 weeks (STAIR/ImRs; WL/ImRs) vs. 36 weeks (WL/STAIR). | baseline and max 36 weeks (depdending on condition)
Post-treatment: Change from Baseline in Inventory of Interpersonal Problems (IIP) at 8 weeks (ImRs) vs 16 weeks (STAIR/ImRs; WL/ImRs) vs. 24 weeks (WL/STAIR). | baseline and max 24 weeks (depending on condition)
12-week FU: Change from Baseline in Inventory of Interpersonal Problems (IIP) at 20 weeks (ImRs) vs 28 weeks (STAIR/ImRs; WL/ImRs) vs. 36 weeks (WL/STAIR). | baseline and max 36 weeks (depdending on condition)
Post-treatment: Change from Baseline in Dissociation Questionnaire (DIS-Q) at 8 weeks (ImRs) vs 16 weeks (STAIR/ImRs; WL/ImRs) vs. 24 weeks (WL/STAIR) | baseline and max 24 weeks (depending on condition)
12-week FU: Change from Baseline in Dissociation Questionnaire (DIS-Q) at 20 weeks (ImRs) vs 28 weeks (STAIR/ImRs; WL/ImRs) vs. 36 weeks (WL/STAIR). | baseline and max 36 weeks (depdending on condition)
Post-treatment: Change from Baseline in WHO-Quality of Life(WHO-QL) at 8 weeks (ImRs) vs 16 weeks (STAIR/ImRs; WL/ImRs) vs. 24 weeks (WL/STAIR) | baseline and max 24 weeks (depending on condition)
12-week FU: Change from Baseline in WHO-Quality of Life(WHO-QL) at 20 weeks (ImRs) vs 28 weeks (STAIR/ImRs; WL/ImRs) vs. 36 weeks (WL/STAIR). | baseline and max 36 weeks (depdending on condition)
Post-treatment: Change from Baseline in Difficulties in Emotion Regulation Scale Post-treatment: Change from Difficulties in Emotion Regulation Scale (DERS) at 8 weeks (ImRs) vs 16 weeks (STAIR/ImRs; WL/ImRs) vs. 24 weeks (WL/STAIR) | baseline and max 24 weeks (depending on condition)
12-week FU: Change from Baseline in Difficulties in Emotion Regulation Scale (DERS) at 20 weeks (ImRs) vs 28 weeks (STAIR/ImRs; WL/ImRs) vs. 36 weeks (WL/STAIR). | baseline and max 36 weeks (depdending on condition)
Post-treatment: Change from Baseline in Structured Clinical Interview - Axis I (SCID-1) at 8 weeks (ImRs) vs 16 weeks (STAIR/ImRs; WL/ImRs) vs. 24 weeks (WL/STAIR) | baseline and max 36 weeks (depdending on condition)
12-week FU: Change from Baseline in Structured Clinical Interview - Axis I (SCID-1) at 20 weeks (ImRs) vs 28 weeks (STAIR/ImRs; WL/ImRs) vs. 36 weeks (WL/STAIR). | baseline and max 36 weeks (depdending on condition)

CONTACTS AND LOCATIONS:
Overall Officials: Merel Kindt, Prof dr, Principal Investigator — University of Amsterdam
Locations (1):
- University of Amsterdam, Amsterdam, Netherlands